CLINICAL TRIAL: NCT03354169
Title: Randomized Controlled Trial Examining the Effects of Meal Timing Among Obese Individuals
Brief Title: Daytime vs. Delayed Eating Among Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kelly Allison, Director, Center for Weight and Eating Disorders, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 828317; R01DK117488 (NIH)
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Obesity
Keywords: Metabolism; Eating; Circadian Rhythms
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Randomized within subjects, cross-over design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Daytime Eating Condition (Experimental): Participants will be asked to eat all of their meals and snacks, as provided by the study, between 0800 and 1900.
  Interventions: Behavioral: Eating Condition
- Delayed Eating Condition (Experimental): Participants will be asked to eat all of their meals and snacks, as provided by the study, between 1200 and 2300.
  Interventions: Behavioral: Eating Condition
- Withdrawn before randomization (Other): Two participants completed the screening process and started the first inpatient assessment visit but were withdrawn prior to completion of the assessment visit and were not randomized to start the intervention. They were not included in data analysis.
  Interventions: Other: No Intervention; withdrawn before randomization

INTERVENTIONS:
Behavioral: Eating Condition — Participants will be randomly assigned to eat per the prescribed eating condition for 8 weeks during eating condition 1. They will complete the alternate eating condition for 8 weeks during eating condition 2.
  Arms: Daytime Eating Condition; Delayed Eating Condition
Other: No Intervention; withdrawn before randomization — These participants were withdrawn and did not receive an intervention.
  Arms: Withdrawn before randomization

SUMMARY:
The randomized, cross-over design study is designed to determine how timing of eating affects weight, adiposity, energy metabolism, and gene expression. Obese participants will be provided isocaloric meals and snacks to be consumed in one of two prescribed eating conditions -- daytime eating and delayed eating.

DETAILED DESCRIPTION:
The study consists of the following phases - screening, assessment visit 1, eating condition 1, assessment visit 2, a wash-out period, assessment visit 3, eating condition 2 and assessment visit 4, as discussed in detail below. The assessment visits will all consist of the same procedures and will take place at the Center for Human Phenomic Science (CHPS) of the Hospital of the University of Pennsylvania before and after each of the eating conditions (four times total). The four 28-hour inpatient assessments will consist of blood draws, adipose (fat) tissue sampling, a dual energy X-ray absorptiometry (DEXA) scan, and a resting metabolic rate test.

During the screening period in order to determine eligibility, participants must complete a 2-part screening visit; This includes:

1. A complete physical examination
2. Tests of blood to screen for any conditions such as diabetes or any serious, uncontrolled medical condition that may interfere with participation in the study.
3. An Electrocardiogram (EKG) test
4. Urine Pregnancy Test
5. Urine Drug Screening
6. the completion of several self-report questionnaires and structured interviews

During the screening period, participants will also be asked to keep a 10-day food log where they will record all food and beverages consumed and their sleep and exercise schedule. Participants will be asked to wear an Actigraph wrist watch at this time.

Following successful completion of the screening period, participants will complete the first of 4 assessment visits. All assessment visits will follow the same protocol.

Assessment Visit Day 1 Procedures:

The visit will include 28 hours (overnight) spent at the CHPS, where meals and snacks will be provided. At each of the assessment visits participants will be given a urine drug screening and, if appropriate, a pregnancy test. The lights will be dim in the hospital room to control for light.

Participants will arrive at 7:00 am. Starting at 8:00 am, blood will be drawn every four hours. From this blood gene expression and hormones related to metabolism, eating, and sleep will be measured.

Following the first blood draw, resting metabolic rate is measured for 45 minutes. Lunch is then provided, followed by a measurement of body composition using a DEXA scan. Next, the adipose tissue sampling procedure will begin. Lastly, the participants will complete a series of cognitive tests administered on a laptop.

Participants will be provided meals and snacks during their visit and are free to watch television or participate in other sedentary pastimes while they are there.

Assessment Visit Day 2 Procedures:

After an overnight fast, participants will undergo the Frequently Sampled Intravenous Glucose Tolerance Test (FSIGT) on the morning of day 2.

Following the FSIGT test, participants will be served a meal and during the first assessment visit, participants will be randomly assigned to start with one of two eating conditions for the next 8 weeks: 1) Daytime or 2) Delayed. Following randomization, participants will be discharged from CHPS and begin eating condition 1.

If participants are assigned to the daytime eating condition first, they will be asked to consume all of their meals and snacks each day between 8:00 am and 7:00 pm. If they are assigned to the delayed eating condition first, they will be asked to consume all of their meals and snacks between 12 noon and 11:00 pm each day. Participants will eat on this schedule for 8 weeks. During the two, 8-week eating periods, all of the meals and snacks will be provided by the research kitchen. During the eating conditions, participants will be asked to complete daily self-report queries concerning their adherence to the food, sleep, and physical activity requirements of the study.

Following eating condition 1, participants will return for assessment visit 2. This assessment visit follows the same procedures as all other assessment visits. Following assessment visit 2, participants will begin their 2 week washout period where they are instructed to eat as they normally would whenever they like. Following the two-week washout period, participants will return for assessment visit 3, after which they will begin eating condition 2. Following 8 weeks of eating condition 2 participants will return for their final visit, assessment visit 4. After this final assessment, participation in the study will be complete.

ELIGIBILITY:
Inclusion Criteria:

* age 21-50
* BMI of 30-50 kg/m2
* stable weight (±10 lb) over the previous 6 months
* women must be pre-menopausal with regular menstrual cycles

Exclusion Criteria:

* unstable, serious medical conditions
* use of medicine linked to weight gain/loss
* cardiac conditions
* cancer
* diabetes
* autoimmune disease
* use of illicit drugs, melatonin, diuretics or hypnotics
* involved in a current weight loss program
* presence of an untreated sleep disorder (determined by surveys and actigraphy)
* those who work shift work
* those with extreme chronotypes
* habitual waking outside of 0600h-0930h
* habitual bedtime <2200h or >2400h
* sleep duration of <6.5 or >8.5 h/night.
* psychiatric exclusions will be: depression (Patient Health Questionnaire-9 score ≥9), lifetime bipolar disorder, psychosis, or eating disorder; or any other severe psychiatric disorder judged to interfere with study adherence as assessed by the MINI International Neuropsychiatric Interview.
* structured exercise >3 d/wk, for >30 min measured by exercise logs and actigraphy; normal activity levels are required during the study (±30 min/wk of baseline level).

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Allison, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Weight and Eating Disorders, Perelman School of Medicine, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Daytime Eating (8 Wks), Followed by Washout (2 Wks), Followed by Delayed Eating (8wks): Participants were asked to eat on the Daytime condition first, eating all of their meals and snacks, as provided by the study, between 0800 and 1900 hr for 8 weeks. They then had a 2-week washout period eating as they liked. Finally, they were on the Delayed condition when they ate their meals between 1200 and 2300 hr for 8 weeks.
- Delayed Eating (8 Wks), Followed by Washout (2 Wks), Followed by Daytime Eating (8wks): Participants were asked to eat on the Delated condition first, eating all of their meals and snacks, as provided by the study, between 1200 and 2300 hr for 8 weeks. They then had a 2-week washout period eating as they liked. Finally, they were on the Daytime condition when they ate their meals between 0800 and 1900 hr for 8 weeks.
Period: Overall Study
Arm/Group | Daytime Eating (8 Wks), Followed by Washout (2 Wks), Followed by Delayed Eating (8wks) | Delayed Eating (8 Wks), Followed by Washout (2 Wks), Followed by Daytime Eating (8wks)
Started | 18 | 18
Completed | 14 | 16
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Population: All study participants are described as they all were intended to complete both eating conditions. Two were withdrawn after their first assessment visit but before randomization occurred.
Groups:
- All Study Participants: Participants will be asked to eat all of their meals and snacks, as provided by the study, between 0800h and 1900h during the Daytime condition and between 1200h and 2300h in the Delayed condition. Participants will be randomly assigned to eat per the prescribed eating condition for 8 weeks during eating condition 1. They will then have a 2-week washout period. They will complete the alternative eating condition for 8 weeks during eating condition 2. Two participants were withdrawn from the study after assessment visit 1 and were not randomized.
Arm/Group | All Study Participants
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.94 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Body Mass (Weight)
Description: changes in body mass, as measured by a calibrated digital scale, will be explored.
Time Frame: pre-post changes between the daytime and delayed eating conditions (each 8 weeks long)
Population: Thirty participants completed the two eating conditions; six were withdrawn prior to completing at least two assessment visits.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Daytime Eating Condition | Delayed Eating Condition
Number analyzed (Participants) | 30 | 30
kg | -2.1067 (3.8373) | -2.1887 (2.7237)

2. Primary Outcome: Adiposity - Total Body Fat
Description: changes in measures of total body fat, as measured by a DEXA scan, will be explored.
Time Frame: pre-post changes between the daytime and delayed eating conditions (8 weeks).
Measure: Mean (Standard Deviation); unit: percentage of total body mass
Arm/Group | Daytime Eating Condition | Delayed Eating Condition
Number analyzed (Participants) | 30 | 30
percentage of total body mass | -0.3300 (1.8217) | -0.4833 (1.2862)

3. Primary Outcome: Energy Homeostasis Outcomes - REE
Description: Changes in resting energy expenditure values will be explored.
Time Frame: pre-post changes between the daytime and delayed eating conditions (8 weeks).
Measure: Mean (Standard Deviation); unit: kcals per day
Arm/Group | Daytime Eating Condition | Delayed Eating Condition
Number analyzed (Participants) | 30 | 30
kcals per day | -32.4723 (260.8070) | 47.0390 (240.9396)

4. Primary Outcome: Energy Homeostasis - Respiratory Quotient
Description: Respiratory quotient (RQ) was measured with a Parvo-Medics metabolic cart. It is calculated from the ratio of carbon dioxide produced by the body to oxygen consumed by the body, when the body is in a steady state.
Time Frame: pre-post changes between the daytime and delayed eating conditions (8 weeks).
Measure: Mean (Standard Deviation); unit: ratio of CO2 produced/O2 consumed
Arm/Group | Daytime Eating Condition | Delayed Eating Condition
Number analyzed (Participants) | 30 | 30
ratio of CO2 produced/O2 consumed | -0.203 (0.0607) | -0.0197 (0.6499)

ADVERSE EVENTS:
Time Frame: We collected adverse event data for up to ~24 weeks, from initial screening visit and consent through the completion of the study for each participant.
Groups:
- Daytime Eating Condition: Adverse events that were experienced during the pre- or post-daytime eating condition inpatient assessment visits are reported in this group.
  No AEs were reported outside of the assessment visits.
- Delayed Eating Condition: Adverse events that were experienced at the pre- or post- Delayed Eating Condition assessment visits are presented in this group.
  No AEs were reported outside of the assessment visits.
- Non-randomized Participants: Two participants experienced adverse events at their first inpatient assessment visits and withdrew from the study. There were not randomized to an eating condition (this occurred at the conclusion of assessment visit 1).
Arm/Group | Daytime Eating Condition | Delayed Eating Condition | Non-randomized Participants
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/2
Other Adverse Events (participants affected / at risk) | 6/36 | 6/36 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daytime Eating Condition (N=36) | Delayed Eating Condition (N=36) | Non-randomized Participants (N=2)
non-infected phlebitis (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 0 (0) — related to FSIGT test
vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
headache (General disorders) | 0 (0) | 2 (2) | 0 (0)
hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) — related to FSIGT test
sub-conjunctive hemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
vein infiltration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — related to FSIGT test
pain in upper left extremity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT03354169/Prot_SAP_001.pdf
  • Informed Consent Form (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT03354169/ICF_000.pdf